CLINICAL TRIAL: NCT05768100
Title: Hemodynamic Effects of Modulating Circulating Ketone Bodies With 1,3-butanediol
Acronym: KETO-BD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-8-23
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — 1,3-butylene glycol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1,3-Butanediol (Experimental)
  Interventions: Dietary Supplement: 1,3-Butanediol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 1,3-Butanediol — 1,3-Butanediol
  Other Names: Ketone-IQ (HVMN)
  Arms: 1,3-Butanediol
Dietary Supplement: Placebo — Isovolumic placebo
  Arms: Placebo

SUMMARY:
Heart Failure (HF) is a major public health issue affecting 1-2% of the Western population and the lifetime risk of HF is 20%. Despite major improvements in the management and care of patients with HF, the 1-year mortality in patients with HF is high. Furthermore, patients with HF have markedly decreased physical capacity and quality of life. Thus, there is a need for new treatment modalities in this group of patients.

In a first-in-man study we have recently discovered that 3-OHB-infusion increases cardiac output by 2 L/min (40% relative increase) and left ventricular (LV) ejection fraction (LVEF) by 8% in absolute numbers in patients with HF and reduced LVEF (HFrEF).

1,3-Butanediol (BD) serves as a potential nutritional supplement in providing long-lasting ketosis as a treatment option in heart disease. Whether BD provides similar hemodynamic effects as ketone monoester remains unknown.

Hypothesis Oral BD increases cardiac output and LV function in patients with HFrEF.

Aims To investigate the acute hemodynamic effects of weight-adjusted oral BD supplements in patients with HFrEF.

Design In a randomized, single-blind, placebo-controlled, crossover design, 12 patients with HFrEF are studied following overnight fast on 2 separate visits in random order: 1) during intake of BD (HVMN, San Francisco, California, USA) and during placebo.

Methods Transthoracic echocardiography, non-invasive blood pressure, and venous blood samples are obtained every 60 minutes from baseline until 6 hours following BD ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HF: NYHA class II-III, LVEF <40%. Negative urine-HCG for women with childbearing potential. Age ≥18 years.

Exclusion Criteria:

* Diabetes or HbA1c >48 mmol/mol, significant cardiac valve disease, severe stable angina pectoris, severe comorbidity as judged by the investigator, inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Cardiac output | 6 hours
  As measured by LVOT VTI and HR

SECONDARY OUTCOMES:
Stroke volume | 6 hours
Heart rate | 6 hours
LVEF | 6 hours
Changes in circulating 3-OHB | 6 hours
Changes in FFA | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Cardiology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guldbrandsen H, Gopalasingam N, Christensen KH, Horsdal OK, Nielsen R, Wiggers H, Berg-Hansen K. Cardiovascular and Metabolic Effects of Modulating Circulating Ketone Bodies With 1,3-Butanediol in Patients With Heart Failure With Reduced Ejection Fraction. J Am Heart Assoc. 2025 Jan 7;14(1):e038461. doi: 10.1161/JAHA.124.038461. Epub 2024 Dec 24. PMID 39719429